CLINICAL TRIAL: NCT00401674
Title: Phase II Multicenter Study of the Combination of Weekly Carboplatin and Paclitaxel as First-line Chemotherapy for Elderly Patients With Ovarian Cancer.
Brief Title: MITO-5: Weekly Carboplatin and Paclitaxel as First Line Chemotherapy for Elderly Patients With Ovarian Cancer
Acronym: MITO-5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITO-5
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; elderly; weekly chemotherapy; first-line
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel

ARMS (1):
- SINGLE ARM (Experimental)
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
The purpose of this study is to evaluate the toxicity and activity of weekly administration of carboplatin and paclitaxel as first-line chemotherapy for elderly patients with ovarian cancer stage IC-IV.

DETAILED DESCRIPTION:
This is a phase II multicenter study. The experimental treatment is carboplatin (AUC 2) and paclitaxel 60 mg/m2, on days 1, 8 and 15 every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or greater
* Cytologic / histologic diagnosis ovarian cancer
* Stage of disease at diagnosis IC -IV
* Performance status (ECOG) < 3
* Indication for chemotherapy treatment
* Written informed consent

Exclusion Criteria:

* Previous or concomitant malignant neoplasia (not including basocellular or spinocellular skin carcinoma or in-situ carcinoma of the uterine cervix, provided they are being adequately treated)
* Cerebral metastases
* Neutrophils < 1000/mm3, platelets < 100000/mm3, hemoglobin < 8g/dl
* Creatinine > o = 1.25 times the upper normal limit
* GOT or GPT > o = 1.25 times the upper normal limit, except in case of liver metastases)
* Patient's inability to comply with followup

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 6 month
Toxicity | up to 6 months
  assessed weekly

SECONDARY OUTCOMES:
possible predictive factors of the geriatric ADL and IADL scales | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples
Locations (10):
- Italy (10):
  - Ospedale Fatebenefratelli, U.O. di Oncologia, Benevento, BN
  - Università Cattolica del Sacro Cuore, Dipartimento di Oncologia, Campobasso, CB
  - Ospedale Cannizzaro, Cannizzaro, CT
  - Azienda Ospedaliera Carlo Poma, Divisione di Oncologia ed Ematologia, Mantova, MN
  - Ospedale S. Massimo, Penne, PE
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma, Roma
  - Ospedale Civile Umberto I, Day Hospital Oncoematologico, Nocera Inferiore, SA
  - Ospedale S. Bortolo ULSS 6, U.O. di Oncologia Medica, Vicenza, VI
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli

REFERENCES:
- [Result] Pignata S, Breda E, Scambia G, Pisano C, Zagonel V, Lorusso D, Greggi S, De Vivo R, Ferrandina G, Gallo C, Perrone F. A phase II study of weekly carboplatin and paclitaxel as first-line treatment of elderly patients with advanced ovarian cancer. A Multicentre Italian Trial in Ovarian cancer (MITO-5) study. Crit Rev Oncol Hematol. 2008 Jun;66(3):229-36. doi: 10.1016/j.critrevonc.2007.12.005. Epub 2008 Feb 1. PMID 18243011